CLINICAL TRIAL: NCT05441579
Title: Application of Behavioral Economic Strategies to Enhance Recruitment Into a Pediatric Randomized Clinical Trial
Brief Title: Recruitment and Behavioral Economic Strategies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed no difference between groups
Sponsor: Vanessa Olbrecht (Other)
Responsible Party: Sponsor-Investigator, Vanessa Olbrecht, Associate Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00002413
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Surgery; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior | interventions — Economics, Behavioral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 - VR-BF BE (Experimental): We are applying Behavioral Economics (BE)-based messaging and presentation strategies to patient recruitment and determining whether these strategies may enhance patient recruitment into a pediatric randomized clinical trial. Phase 1 will focus on patients that would be enrolled into a biofeedback-based virtual reality (VR-BF) arm.
  Interventions: Behavioral: Behavioral Economics (BE) recruitment strategies; Other: Biofeedback-based virtual reality (VR-BF)
- Phase 1 - VR-BF Biological (Active Comparator): A similar to BE-based recruitment video using a standard biological approach on teenagers' decision to enroll in a clinical study will be used as comparison. Phase 1 will focus on patients that would be enrolled into a biofeedback-based virtual reality (VR-BF) arm.
  Interventions: Other: Biofeedback-based virtual reality (VR-BF)
- Phase 2 - Manage My Pain BE (Experimental): We are applying Behavioral Economics (BE)-based messaging and presentation strategies to patient recruitment and determining whether these strategies may enhance patient recruitment into a pediatric randomized clinical trial. Phase 2 will focus on patients that would be enrolled into the control arm of a clinical trial with a control intervention, Manage My Pain application.
  Interventions: Behavioral: Behavioral Economics (BE) recruitment strategies; Other: Manage My Pain
- Phase 2 - Manage My Pain Biological (Placebo Comparator): A similar to BE-based recruitment video using a standard biological approach on teenagers' decision to enroll in a clinical study will be used as comparison. Phase 2 will focus on patients that would be enrolled into the control arm of a clinical trial with a control intervention, Manage My Pain application.
  Interventions: Other: Manage My Pain

INTERVENTIONS:
Behavioral: Behavioral Economics (BE) recruitment strategies — Behavioral economics (BE), a method of economic analysis that applies psychological insights into human behavior to explain economic decision-making, has broad applicability and its techniques offer a novel way that may be applied to try to help enhance study recruitment and enrollment.
  Arms: Phase 1 - VR-BF BE; Phase 2 - Manage My Pain BE
Other: Biofeedback-based virtual reality (VR-BF) — Phase 1 will focus on patients that would be enrolled into a biofeedback-based virtual reality (VR-BF) arm.
  Arms: Phase 1 - VR-BF BE; Phase 1 - VR-BF Biological
Other: Manage My Pain — Commercially available and free app to track, analyze and monitor pain.
  Arms: Phase 2 - Manage My Pain BE; Phase 2 - Manage My Pain Biological

SUMMARY:
To determine the impact of the application of behavioral economic strategies on recruitment of pediatric patients into a randomized clinical trial assessing the impact of technology-based interventions on postoperative pain management.

DETAILED DESCRIPTION:
Patients will be asked to watch one of two videos in either Phase 1 or Phase 2 relating to recruitment and fill out a survey to determine their likelihood to enroll in a research study. Patients 12-18 years of age presenting for surgery that requires postoperative admission and usually requires narcotic administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 12-18 years of age
* Patients able to read, understand, and speak English
* Patients undergoing surgery requiring postoperative admission
* Patients undergoing surgery that requires narcotic administration

Exclusion Criteria:

* Patients outside of the age range
* Patients with history of developmental delay, uncontrolled psychiatric conditions, or neurological conditions (i.e., epilepsy, motion sickness, nausea/vomiting)
* History of severe vertigo or dizziness
* History of chronic pain
* Patients that use opioids or benzodiazepines chronically
* Patients with conditions that would preclude placement of a VR headset, including craniofacial abnormalities or undergoing surgeries of the head and neck.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 2 was not initiated and was discontinued due to statistical futility.
Groups:
- Phase 2 - Manage My Pain BE: Control arm of trial with the control intervention, Manage My Pain application with a script and film using a BE-informed recruitment video.
- Phase 2 - Manage My Pain Biological: Control arm of trial with the control intervention, Manage My Pain application with a script and film using a recruitment video using a standard biological approach.
Period: Overall Study
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological | Phase 2 - Manage My Pain BE | Phase 2 - Manage My Pain Biological
Started | 64 | 64 | 0 | 0
Completed | 64 | 64 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.6) | 14.6 (1.6) | 14.7 (1.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 31 | 33 | 64
  Female | 32 | 31 | 63
  Prefer not to answer | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 60 | 61 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 50 | 53 | 103
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 64 | 64 | 128
Previous pain management [Count of Participants; unit: Participants] — Type of pain management used in the past.
  Participants
    Over-the-counter pain medication | 59 | 58 | 117
    Massage | 7 | 13 | 20
    Acupuncture | 1 | 1 | 2
    Chiropractor | 6 | 4 | 10
    Prescribed pain medication | 13 | 20 | 33
    Deep breathing, meditation, guided imagery, relaxation or similar approach | 9 | 16 | 25
    Have not had pain in the past | 0 | 0 | 0
    Other | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Impact of the Application of Behavioral Economic Strategies on Recruitment of Pediatric Patients Into a Randomized Clinical Trial Assessing the Impact of Technology-based Interventions on Postoperative Pain Management.
Description: Survey to identify likelihood to participate in study using a 5-point Likert scale (1="Extremely Unlikely" to 5="Extremely Likely").
Time Frame: Baseline
Population: Two participants from the standard recruitment video group did not respond to questions related to this outcome.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 62
score on a scale
  Interest in using ForeVR | 4 [3 to 4] | 4 [3 to 4]
  Interest in participating in clinical trial involving ForeVR | 3 [3 to 4] | 4 [3 to 4]

2. Primary Outcome: Willingness to Participate in Clinical Trial
Description: If given the opportunity, would you participate in the clinical trial?
Time Frame: Baseline
Population: Two participants from the standard recruitment video group did not respond to questions related to this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 62
Participants
  Yes | 48 | 49
  No | 16 | 13

3. Secondary Outcome: Intention to Adhere to Therapy - Would Practice
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I would practice this technology at least once per day before surgery.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 4 [3 to 4] | 4 [3 to 4]

4. Secondary Outcome: Acceptability of Therapy - Excitement
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I would be excited to use this technology.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 4 [3 to 4] | 4 [3 to 4]

5. Secondary Outcome: Perception of Efficacy - Less Pain
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I believe this technology would help me have less pain after surgery.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 3 [3 to 4] | 3 [3 to 4]

6. Secondary Outcome: Perception of Risk - Side Effects
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I am worried that this technology would have a lot of side effects.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 2 [1 to 2] | 2 [2 to 3]

7. Secondary Outcome: Opinion of Treatment Burden - Ease of Use
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I feel that this technology would be easy to use.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 3 [3 to 4] | 4 [3 to 4]

8. Secondary Outcome: Intention to Adhere to Therapy - Would Use
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I would use this technology at least once per day after surgery while I was still needing it.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 4 [3 to 4] | 4 [3 to 4]

9. Secondary Outcome: Acceptability of Therapy - Pain Medication
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I would like to use this technology to help me take less pain medication.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 4 [3 to 4] | 4 [3 to 4]

10. Secondary Outcome: Acceptability of Therapy - Recommend to Others
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I would recommend this therapy to other individuals undergoing surgery.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 4 [3 to 4] | 4 [3 to 4]

11. Secondary Outcome: Acceptability of Therapy - Preference
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I would prefer using this technology over taking pain medications.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 4 [3 to 4] | 4 [3 to 4]

12. Secondary Outcome: Perception of Efficacy - Less Pain Medication
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I believe that this technology would help me use less pain medication after surgery.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 3 [3 to 4] | 3 [3 to 4]

13. Secondary Outcome: Perception of Risk - Amount
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I believe that this technology would be too risky for me to use.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 2 [1 to 2] | 2 [2 to 3]

14. Secondary Outcome: Opinion of Treatment Burden - Independence
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I would feel comfortable using this technology independently without supervision.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 3 [3 to 4] | 4 [3 to 4]

15. Secondary Outcome: Opinion of Treatment Burden - Familiar
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I am familiar with how to use this type of technology.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 3 [3 to 4] | 4 [3 to 4]

16. Secondary Outcome: Opinion of Treatment Burden - Pay for Technology
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I would pay for the opportunity to use this technology during my recovery.
  I am comfortably using technologies like this.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 3 [3 to 4] | 4 [3 to 4]

17. Secondary Outcome: Opinion of Treatment Burden - Technology Comfort
Description: Based on answers to the following survey questions which were assessed along a 5-point Likert scale (from 1="Strongly Disagree" to 5= "Strongly Agree"):
  I am comfortably using technologies like this.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a Likert scale
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
Number analyzed (Participants) | 64 | 64
score on a Likert scale | 3 [3 to 4] | 4 [3 to 4]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Phase 1 - VR-BF BE | Phase 1 - VR-BF Biological
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT05441579/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT05441579/SAP_001.pdf